

## **Specialized Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Project PISCES I: Precision Implemented Smoking Cessation Evaluation Study 2019-0953

**Subtitle: PISCES Questionnaire Statement** 

Study Chair: Jason Robinson

## Goal of the Study:

- To find out how to personalize treatments for quitting smoking based on unique character traits
- To potentially help doctors individualize smoking cessation treatment for people who do not quit smoking after an initial course of treatment
- The study is divided into two six-week stages (total of twelve weeks of treatment) followed by 3 month and 6 month follow up visits.

## Requirements to Proceed with Screening Process:

- You will electronically sign an informed consent document at your upcoming baseline screening phone visit.
- In preparation for your screening phone visit, you will complete the attached questionnaires. This will decrease the time needed to complete the phone visit.

### Purpose of This Questionnaire Consent:

 So that you may complete the screening questionnaires prior to signing the screening consent form.

### About the Questionnaires:

- The questionnaires attached will ask you about depression, emotions, motivation, negative events and your dependence on smoking.
- The questionnaires should take less than 45 minutes to complete.

#### **Questionnaire Consent Statement**

I have read the description of the study and agree to answer all questionnaires associated with screening and enrollment (if I am eligible to be enrolled). I understand that I may refuse to answer any (or all) of the questions and may refuse study participation. I understand that I must complete the questionnaires before the study phone call, or I may not be able to participate.

During the course of this study, the research team at The University of Texas MD Anderson Cancer Center will be collecting information about me that they may share with health authorities and study monitors. By answering the questions, I am providing authorization for the research team to use and share my information at any time. There is no expiration date for the use of this information. I may withdraw my authorization at any time, in writing, for any reason. I may contact PISCES staff with any questions at (713) 792-2265.

-----

[Participant will then see the Questionnaires Link here]